CLINICAL TRIAL: NCT07007182
Title: A Randomized, Controlled, Multicenter Phase II Study of Conversion Therapy Combined With Surgery and Radiotherapy for Retroperitoneal Lymph Node Metastases in Gastric Cancer
Brief Title: Conversion Therapy Plus Surgery and Radiotherapy for Retroperitoneal Nodal Metastases in Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinbo Yue (Other)
Responsible Party: Sponsor-Investigator, Jinbo Yue, Professor of Radiation Oncology; Principal Investigator, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-150-02
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Gastric Adenocarcinoma; Stomach Neoplasms
Keywords: Conversion therapy; Para-aortic lymph nodes; D2 gastrectomy; Radiotherapy; SOX regimen; Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; S 1 (combination); Tegafur; XELOX; Capecitabine; Immune Checkpoint Inhibitors; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversion therapy + surgery + para-aortic radiotherapy (Experimental): Patients with isolated para-aortic (station 16) lymph node metastases from gastric adenocarcinoma will receive first-line systemic conversion therapy based on PD-L1 combined positive score (CPS).
  * CPS ≥1: 3 cycles of SOX (S-1 plus oxaliplatin) plus a PD-1 inhibitor (every 3 weeks).
  * CPS <1: 3 cycles of SOX alone. After ~8 weeks, patients with non-progressive disease (CR/PR/SD) undergo D2 radical gastrectomy, followed by 5 cycles of adjuvant SOX.
  Subsequently, patients receive elective intensity-modulated radiotherapy (IMRT) to the para-aortic (station 16) nodal basin (45-50 Gy/25 fractions; positive nodes 56-60 Gy/25 fractions) with concurrent oral capecitabine or S-1.
  For CPS ≥1 patients, maintenance PD-1 inhibitor therapy continues for up to 1 year.
  Interventions: Drug: SOX regimen; Drug: PD-1 inhibitor; Radiation: Para-aortic lymph node radiotherapy (IMRT to station 16); Drug: Capecitabine / S-1 (radiosensitizer during IMRT)
- Systemic therapy alone (Active Comparator): Patients in this arm will receive systemic therapy without surgery or radiotherapy.
  * CPS ≥1: CAPEOX or SOX chemotherapy combined with a PD-1 inhibitor, followed by PD-1 inhibitor maintenance for up to 1 year.
  * CPS <1: CAPEOX or SOX chemotherapy alone. Systemic therapy continues until disease progression, unacceptable toxicity, or completion of 8 planned cycles.
  Interventions: Drug: SOX regimen; Drug: CAPEOX regimen; Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: SOX regimen — The SOX regimen consists of oxaliplatin 130 mg/m² IV on day 1 plus oral S-1 (tegafur/gimeracil/oteracil) 40-60 mg twice daily, taken on days 1-14 followed by 7 days off, in a 21-day cycle.
  Experimental arm: 3 cycles before surgery, 5 cycles after surgery. Control arm: up to 8 cycles as standard systemic therapy.
  Other Names: Oxaliplatin + S-1 (tegafur/gimeracil/oteracil)
Drug: CAPEOX regimen — The CAPEOX regimen consists of oxaliplatin 130 mg/m² IV on day 1 plus oral capecitabine 1000 mg/m² twice daily on days 1-14, repeated every 3 weeks (q3w), up to 8 cycles.
  Used as a standard chemotherapy option in the control arm, with or without PD-1 inhibitor according to PD-L1 CPS score.
  Other Names: Oxaliplatin + Capecitabine
  Arms: Systemic therapy alone
Drug: PD-1 inhibitor — A PD-1 inhibitor is administered intravenously at a fixed dose of 200 mg every 3 weeks.
  It is combined with SOX in the experimental arm (CPS ≥1 patients) during conversion and adjuvant phases, and with CAPEOX or SOX in the control arm (CPS ≥1 patients).
  Maintenance PD-1 inhibitor continues for up to 1 year or until disease progression or unacceptable toxicity.
  Other Names: Anti-PD-1 antibody
Radiation: Para-aortic lymph node radiotherapy (IMRT to station 16) — Intensity-modulated radiotherapy (IMRT) is delivered postoperatively to the para-aortic (station 16) nodal basin.
  Elective nodal basin: 45-50 Gy in 25 fractions Positive nodes: 56-60 Gy in 25 fractions Radiotherapy is given concurrently with oral capecitabine or S-1 as radiosensitizers.
  Other Names: IMRT to station 16
  Arms: Conversion therapy + surgery + para-aortic radiotherapy
Drug: Capecitabine / S-1 (radiosensitizer during IMRT) — During para-aortic IMRT, patients receive concurrent oral capecitabine 825 mg/m² twice daily on radiation days, or oral S-1 dosed according to body surface area.
  These agents are used as radiosensitizers during postoperative radiotherapy.
  Other Names: Capecitabine (Xeloda), S-1 (tegafur/gimeracil/oteracil)
  Arms: Conversion therapy + surgery + para-aortic radiotherapy

SUMMARY:
This is a randomized, controlled, multicenter phase II clinical trial evaluating the efficacy and safety of conversion therapy combined with radical gastrectomy and adjuvant radiotherapy targeting para-aortic (station 16) lymph nodes in patients with gastric adenocarcinoma and isolated station 16 nodal metastases. Eligible participants must have no evidence of peritoneal dissemination, visceral metastases, or non-regional lymphatic spread. Based on PD-L1 combined positive score (CPS), patients in the experimental arm will receive systemic therapy with SOX (S-1 plus oxaliplatin) with or without a PD-1 inhibitor, followed by D2 gastrectomy and postoperative adjuvant SOX chemotherapy, then intensity-modulated radiotherapy (IMRT) to the para-aortic region. The control arm will receive standard chemotherapy with CAPEOX or SOX, with or without immunotherapy, according to CPS status. The primary endpoint is progression-free survival (PFS), with secondary endpoints including overall survival (OS), objective response rate (ORR), disease control rate (DCR), and safety. This study aims to explore whether the addition of locoregional treatment to systemic therapy improves long-term outcomes in this select patient population.

DETAILED DESCRIPTION:
This study targets patients with gastric adenocarcinoma characterized by a low metastatic burden-specifically, isolated metastases to para-aortic (station 16) lymph nodes without evidence of peritoneal carcinomatosis, distant organ metastases, or non-regional lymph node involvement. Patients are stratified by PD-L1 combined positive score (CPS ≥1 vs. <1) and receive first-line systemic conversion therapy with the SOX regimen (S-1 plus oxaliplatin), with or without a PD-1 inhibitor. In the experimental arm, patients demonstrating disease control (CR/PR/SD) undergo D2 radical gastrectomy, followed by five cycles of adjuvant SOX and intensity-modulated radiotherapy (IMRT) targeting the station 16 nodal basin (45-50 Gy/25 fractions; positive nodes 56-60 Gy/25 fractions), with concurrent capecitabine or S-1. Maintenance immunotherapy continues for up to one year in CPS ≥1 patients. The control arm receives standard-of-care systemic treatment with CAPEOX or SOX ± immunotherapy, without surgery or radiotherapy. Tumor tissue, peripheral blood, and fecal samples will be collected at multiple time points for exploratory biomarker analyses, including tumor immune microenvironment profiling, tumor mutational burden (TMB), mismatch repair status (MSI), and circulating immune cell subsets. A total of 54 patients will be enrolled (2:1 randomization), with an accrual period of 18 months and 24 months of follow-up.

ELIGIBILITY:
Inclusion:

Histologically confirmed gastric adenocarcinoma with isolated para-aortic (station 16) lymph node metastasis; pMMR or MSS subtype; ECOG performance status 0-2; Life expectancy ≥ 3 months; Adequate organ function (hematologic, hepatic, renal); Ability to provide tumor tissue for biomarker analysis; Ability to understand and willingness to sign written informed consent; Women of childbearing potential must have a negative pregnancy test and agree to use effective contraception during study and for 12 months after treatment; men with partners of childbearing potential must also agree to contraception.

Exclusion Criteria:

Evidence of visceral or peritoneal metastasis; MSI-H or dMMR subtype; HER2-positive disease (IHC 3+ or IHC 2+ with FISH positive); Prior systemic anti-tumor therapy; Prior malignancy within 3 years (except adequately treated basal cell/squamous cell carcinoma of the skin or in situ carcinoma); Prior PD-1/PD-L1/CTLA-4 therapy; Participation in another interventional trial within 4 weeks; Active autoimmune disease requiring systemic therapy within past 2 years; Uncontrolled infection, hepatitis B, C, or HIV; CNS metastases or carcinomatous meningitis; Uncontrolled cardiovascular disease (unstable angina, recent MI, NYHA III-IV heart failure, QTc ≥480 ms); Interstitial lung disease or uncontrolled pulmonary disease; Uncontrolled diabetes mellitus (FBG >10 mmol/L); Pregnancy or breastfeeding; Major surgery within 4 weeks prior to randomization; Any other condition that may interfere with protocol compliance or increase risk as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Time from randomization to disease progression according to RECIST 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  Time from randomization to death from any cause.
Objective Response Rate (ORR) | Up to 6 months after randomization
  Proportion of patients achieving complete or partial response according to RECIST 1.1.
Disease Control Rate (DCR) | Up to 6 months after randomization
  Proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.
Adverse Events (Safety Profile) | Through study completion (approx. 3 years)
  Incidence and grade of treatment-related adverse events according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, MD, PhD, Principal Investigator — Shandong Cancer Hospital and Institute; Jie Chai, MD, PhD, Study Chair — Shandong Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: No